CLINICAL TRIAL: NCT06404112
Title: RECOVER-SLEEP: A Platform Protocol for Evaluation of Interventions for Sleep Disturbances in Post-Acute Sequelae of SARS-CoV-2 Infection (PASC)
Brief Title: RECOVER-SLEEP: Platform Protocol, Appendix_B (CPSD)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00112484_B; OTA-21-015G (Other Grant/Funding Number: NIH Grant to RTI; RTI subcontracting with DCRI)
Record Dates: First submitted 2024-05-06; First posted 2024-05-08 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Long COVID; Long COVID-19; Sleep Disturbance
Keywords: PASC; Sleep Disturbances
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Parasomnias | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: This platform protocol is designed to allocate participants into an intervention appendix based on their symptoms of sleep disturbance. Within the appendix, participants will be randomly assigned based on the appendix study design. Site investigators and personnel will be informed as to which study intervention appendix participants are assigned, but they will be blinded to whether participants are receiving the active study intervention or control, when possible. Similarly, participants will be blinded to active intervention or control, when possible. Randomization will be stratified by the study site; other stratification factors may be considered per appendix.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Active TL + Oral Melatonin (Active Comparator): The Complex PASC-Related Sleep Disturbances (CPSD) Appendix B combines brief education and a tailored sleep timing prescription for CPSD (referred to as RESET-PASC) with therapies that modify circadian timing for participants who report poor sleep quality. The intervention therapies involve tailored lighting (TL) and melatonin. Participants will be randomly assigned to one of four groups: (a) active TL + oral melatonin, (b) active TL + placebo melatonin, (c) placebo TL + oral melatonin, and (d) placebo TL + placebo melatonin. All groups will receive RESET-PASC. The intervention duration will be 8 weeks.
  Interventions: Drug: Melatonin; Device: Tailored lighting (TL) Active
- Active TL + Placebo Melatonin (Active Comparator): The Complex PASC-Related Sleep Disturbances (CPSD) Appendix B combines brief education and a tailored sleep timing prescription for CPSD (referred to as RESET-PASC) with therapies that modify circadian timing for participants who report poor sleep quality. The intervention therapies involve tailored lighting (TL) and melatonin. Participants will be randomly assigned to one of four groups: (a) active TL + oral melatonin, (b) active TL + placebo melatonin, (c) placebo TL + oral melatonin, and (d) placebo TL + placebo melatonin. All groups will receive RESET-PASC. The intervention duration will be 8 weeks.
  Interventions: Drug: Melantonin Placebo; Device: Tailored lighting (TL) Active
- Placebo TL + Oral Melatonin (Active Comparator): The Complex PASC-Related Sleep Disturbances (CPSD) Appendix B combines brief education and a tailored sleep timing prescription for CPSD (referred to as RESET-PASC) with therapies that modify circadian timing for participants who report poor sleep quality. The intervention therapies involve tailored lighting (TL) and melatonin. Participants will be randomly assigned to one of four groups: (a) active TL + oral melatonin, (b) active TL + placebo melatonin, (c) placebo TL + oral melatonin, and (d) placebo TL + placebo melatonin. All groups will receive RESET-PASC. The intervention duration will be 8 weeks.
  Interventions: Drug: Melatonin; Device: Tailored lighting (TL) Placebo
- Placebo TL + Placebo Melatonin (Placebo Comparator): The Complex PASC-Related Sleep Disturbances (CPSD) Appendix B combines brief education and a tailored sleep timing prescription for CPSD (referred to as RESET-PASC) with therapies that modify circadian timing for participants who report poor sleep quality. The intervention therapies involve tailored lighting (TL) and melatonin. Participants will be randomly assigned to one of four groups: (a) active TL + oral melatonin, (b) active TL + placebo melatonin, (c) placebo TL + oral melatonin, and (d) placebo TL + placebo melatonin. All groups will receive RESET-PASC. The intervention duration will be 8 weeks.
  Interventions: Drug: Melantonin Placebo; Device: Tailored lighting (TL) Placebo

INTERVENTIONS:
Drug: Melatonin — Melatonin dosing will be one tablet of 3 mg immediate release daily consumed 2 hours before the participant's desired bedtime, which is defined as the time at which the participant tries to fall asleep.
  Arms: Active TL + Oral Melatonin; Placebo TL + Oral Melatonin
Drug: Melantonin Placebo — Melatonin placebo dosing will be one placebo tablet once daily consumed 2 hours before the participant's desired bedtime.
  Arms: Active TL + Placebo Melatonin; Placebo TL + Placebo Melatonin
Device: Tailored lighting (TL) Active — TL will be delivered similarly to both active and placebo groups, but the circadian stimulus (the amount of light) will be different, albeit practically unidentifiable to participants.
  Arms: Active TL + Oral Melatonin; Active TL + Placebo Melatonin
Device: Tailored lighting (TL) Placebo — TL will be delivered similarly to both active and placebo groups, but the circadian stimulus (the amount of light) will be different, albeit practically unidentifiable to participants.
  Arms: Placebo TL + Oral Melatonin; Placebo TL + Placebo Melatonin

SUMMARY:
The platform protocol is designed to be flexible so that it is suitable for a range of study settings and intervention types. Therefore, the platform protocol provides a general protocol structure that can be shared by multiple interventions and allows comparative analysis across the interventions. For example, objectives, measures, and endpoints are generalized in the platform protocol, but intervention-specific features are detailed in separate appendices.

This platform protocol is a prospective, multi-center, multi-arm, randomized controlled platform trial evaluating potential interventions for PASC-mediated sleep disturbances. The hypothesis is that symptoms of sleep and circadian disorders that emerge in patients with PASC can be improved by phenotype-targeted interventions. Specific sleep and circadian disorders addressed in this protocol include sleep-related daytime impairment (referred to as hypersomnia) and complex PASC-related sleep disturbance (reflecting symptoms of insomnia and sleep-wake rhythm disturbance).

DETAILED DESCRIPTION:
Interventions will be added to the platform protocol as appendices. Each appendix will leverage all elements of the platform protocol, with additional elements described in the individual appendix.

After completing Baseline assessments, participants will be randomized to an intervention group, which is based on their sleep phenotype, or into a placebo/control group.

ELIGIBILITY:
Inclusion Criteria:

• See NCT06404086 for RECOVER-SLEEP: Platform Protocol level inclusion criteria which applies to this appendix

Exclusion Criteria:

• See NCT06404086 for RECOVER-SLEEP: Platform Protocol level exclusion criteria which applies to this appendix

Additional Appendix B (CPSD) Level Inclusion Criteria:

The following additional exclusion criteria are to be considered together for determining eligibility. They are separated here by TL and melatonin only for presentation. RESET-PASC presents no additional exclusions.

TAILORED LIGHTING EXCLUSION CRITERIA

1. Severe visual impairments affecting sensitivity or ability to respond to light
2. Severe photosensitivity dermatitis
3. Severe progressive retinal disease, eg, macular degeneration
4. Permanently dilated pupil, eg, following certain cataract surgeries
5. Unwilling to remove or not wear blue-light-blocking glasses during TL dosing

MELATONIN EXCLUSION CRITERIA

1. Sleep medication, if not willing to washout for 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Change in total score of the PROMIS 8b SD to assess sleep disturbance | Baseline, End of Intervention (Day 63)
  The PROMIS 8b SD form includes a total of 8 items that ask participants to reflect on their sleep over the past 7 days with one question rated very poor to very good and the remaining questions rated not at all to very much. T-Scores range from 0 to 100, with a score of 55 being 1 standard deviation above population mean. Higher scores indicate more sleep disturbance.
Change in sleep onset variability, assessed using a wearable device | Baseline, End of Intervention (Day 63)
  A wearable device will be used as an objective measure to assess sleep onset variability assessed for 7 days before randomization and 7 days before EOI

SECONDARY OUTCOMES:
Change in total score of the PROMIS 8a SRI to assess sleep-related impairment | Baseline, End of Intervention (Day 63)
  The PROMIS 8a SRI form includes a total of 8 items that ask participants to reflect on their sleep-related daytime impairment over the past 7 days with questions rated not at all to very much. T-Scores range from 0 to 100, with > 55 1 SD above population mean.
Change in PROMIS 10a Fatigue score | Baseline, End of Intervention (Day 63)
  The PROMIS 10a Fatigue is a 10-item questionnaire that assesses a participant's fatigue on a scale of 1 (not at all fatigued) to 5 (very much).
Change in an objective neurocognitive battery score | Baseline, End of Intervention (Day 63)
Change in ECog2 measure | Baseline, End of Intervention (Day 63)
  Everyday Cognition 2 (ECog2) is a self-report, 41-item questionnaire used to measure measure the participant's perceived capacity to perform activities related to cognitive function, which could impact major activities of daily living and independence. It has been used for patients with mild cognitive impairment, Alzheimer's Disease, and dementia. It takes 5 minutes to complete.
Change in PASC Symptom Questionnaire responses | Baseline, End of Intervention (Day 63)
  Participants will be asked to complete a questionnaire that asks about the presence of PASC symptoms at Baseline and at follow-up visits. This questionnaire includes symptoms that have been associated with PASC.
Change in total score from ISI (Insomnia Severity Index) | Baseline, End of Intervention (Day 63)
  The ISI is a 7-item, self-report questionnaire that assesses the nature, severity, and impact of insomnia, on a 5-point Likert scale (eg, 0 = not at all, 4 = extremely; scores: from 0 to 28). The ISI asks patients to recall their insomnia symptoms over the past 2 weeks.
Change in within-person variability (over a 7-day period) in sleep onset time, assessed by sleep diary | Baseline, End of Intervention (Day 63)
  Sleep onset time will be assessed by sleep diary
Change in average (over a 7-day period) nocturnal sleep duration, assessed by sleep diary | Baseline, End of Intervention (Day 63)
  Nocturnal sleep duration will be assessed by sleep diary
Change in average (over a 7-day period) 24-hour sleep duration, assessed by sleep diary | Baseline, End of Intervention (Day 63)
  24-hour sleep duration will be assessed by sleep diary
Change in average (over a 7-day period) sleep midpoint, assessed by sleep diary | Baseline, End of Intervention (Day 63)
  Sleep midpoint is the time half way between start and end of sleep, as assessed by sleep diary
Change in average (over a 7-day period) nocturnal sleep duration, assessed by activity tracker | Baseline, End of Intervention (Day 63)
  Nocturnal sleep duration will be assessed by activity tracker
Change in average (over a 7-day period) 24-hour sleep duration, assessed by activity tracker | Baseline, End of Intervention (Day 63)
  24-hour sleep duration will be assessed by activity tracker
Change in average (over a 7-day period) sleep efficiency, assessed by activity tracker | Baseline, End of Intervention (Day 63)
  Sleep Efficiency is the percentage of the sleep period spent asleep, as measured by activity tracker
Change in average (over a 7-day period) sleep midpoint, assessed by activity tracker | Baseline, End of Intervention (Day 63)
  Sleep midpoint is the time half way between start and end of sleep, as assessed by sleep diary

CONTACTS AND LOCATIONS:
Overall Officials: Christina Barkauskas, MD, Study Chair — Duke Clinical Research Institute; Susan Redline, MD MPH, Study Chair — Brigham and Women's Hospital
Locations (1):
- All sites listed under NCT06404086, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The summary of results will be shared on the study website: https://recovercovid.org/

REFERENCES:
- See also: Related Info — http://recovercovid.org/

DOCUMENTS (1):
  • Informed Consent Form (2025-01-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT06404112/ICF_000.pdf